CLINICAL TRIAL: NCT01718730
Title: Cortical Excitability and Inhibition in Children and Adolescents With Major Depressive Disorder
Brief Title: Cortical Excitability and Inhibition in MDD
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Principal Investigator, Paul E. Croarkin, PI, Mayo Clinic
Other Study IDs: 12-000335; NCT00896090 (obsolete NCT alias)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder, Recurrent, Mild; Depressive Disorder, Major
Keywords: TMS; Adolescent; Child; MDD; Major depressive disorder; Mild MDD; Mild depression; SSRI; Motor cortex; Cortical excitability; Cortical inhibition; Cortical silent period; Motor threshold; Intracortical facilitation; Intracortical inhibition; gamma-aminobutyric acid (GABA); Glutamate; N-methyl-D-aspartate (NMDA); Magnetic resonance spectroscopy; MRS
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Lymphoma, Follicular | interventions — Transcranial Magnetic Stimulation; Magnetic Resonance Spectroscopy; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (4):
- Mild depression: Subjects with mild, but clinically significant depression
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Magnetic Resonance Spectroscopy and Imaging
- Moderate to Severe MDD: Subjects with moderate to severe major depressive disorder who have not yet initiated treatment with an SSRI
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Magnetic Resonance Spectroscopy and Imaging
- MDD with response to SSRI: Subjects with moderate to severe major depressive disorder that has responded to an SSRI
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Magnetic Resonance Spectroscopy and Imaging
- MDD without response to SSRI: Subjects with moderate to severe major depressive disorder which has not responded to treatment with an SSRI
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Magnetic Resonance Spectroscopy and Imaging

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Single and paired-pulse TMS applied to the motor cortex will collect measures of cortical excitability and inhibition.
  Other Names: Device: Magstim Model 200
Device: Magnetic Resonance Spectroscopy and Imaging — MRS/MRI Scans will examine glutamate concentrations in the motor cortex and anterior cingulate cortex.
  Other Names: MRS/MRI

SUMMARY:
The purpose of this study is to learn if measures of brain activity are different in children and adolescents with depression who are in different stages of treatment. This is important because it may identify a biological marker for depression that could one day be used to identify depressed children who would benefit from certain treatments (medications for example), or to monitor how well treatments are working. Brain activity measures(known as cortical excitability and inhibition) will be collected by Transcranial Magnetic Stimulation (TMS). TMS is a noninvasive (no surgery or implants) brain stimulation technology which can make parts of the brain work without putting any wires or chemicals into the body. Measurements will take place over one 3-hour visit. This study does not provide any form of treatment.

*There is an optional portion of the study that uses a brain scan to gather measures of brain structure and brain chemicals. The brain scan is called magnetic resonance and spectroscopy (MRI/MRS). MRI/MRS uses magnetic fields to study the structure of the brain and brain chemicals. The PI will determine eligibility for the MRI/MRS portion of the study.

DETAILED DESCRIPTION:
This study is focused on understanding the neurophysiology of major depressive disorder (MDD), and the impact of selective serotonin reuptake inhibitors (SSRIs) in children and adolescents. This is a cross-sectional study which will utilize single and paired-pulse transcranial magnetic stimulation (TMS) to collect measures of glutamatergic cortical excitability (the motor threshold and intracortical facilitation), and GABAergic cortical inhibition (the cortical silent period and intracortical inhibition) of the motor cortex in chilren and adolescents in various disease states of MDD. The optional proton magnetic resonance spectroscopy and imaging scans (MRS/MRI) at 3 Tesla (3T) will examine glutamate concentrations in the motor cortex and anterior cingulate cortex.

This is a biomarker study (MRI/MRS and TMS neurophysiology measures); treatment is not provided in any form. This study will not utilize Repetitive Transcranial Magnetic Stimulation (rTMS).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents from the ages of 13 to 21, male or female.
* Subjects with MDD (groups 2, 3, and 4):
* Must have a Children's Depression Rating Scale, Revised (CDRS-R) score of 40 or higher
* Must have a Clinical Global Impression-Severity scale (CGI-S) score of 4 or higher.
* Group 1: (50 subjects): Subjects who have mild (CDRS-R score < 40) but clinically significant depression.
* Group 2: (50 subjects): Subjects with moderate to severe MDD who have not yet initiated treatment with an SSRI.
* Group 3: (50 subjects): Subjects with moderate to severe MDD that has responded to treatment with an SSRI.
* Group 4: (50 subjects): Subjects with moderate to severe MDD which has not responded to treatment with an SSRI.
* Capable of providing informed assent (consent if age 18) in addition to consent by parent or guardian.
* Subjects and at least 1 parent must be fluent in English.

Exclusion Criteria:

* Primary Axis I or II disorder other than MDD.
* Unprovoked seizure history, seizure disorder, history of febrile seizures, family history of epilepsy.
* Any significant findings on the TMS Adult Safety Screen (TASS) or contraindications to MRI/MRS
* Subjects who are judged by the Principal Investigator to be at imminent risk for self harm or suicide as indicated by interview or C-SSRS.
* Pregnancy or suspected pregnancy in females.
* Metal in the head (except the mouth*), implanted medication pumps, cardiac pacemaker.

  * Subjects with braces will be excluded from MRI/MRS portion of study only
* Prior brain surgery.
* Risk for increased intracranial pressure such as a brain tumor.
* Any unstable medical condition.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This protocol will plan to screen depressed children and adolescents who are seeking treatment at Mayo Clinic in Rochester, MN, using strict inclusion and exclusion criteria. These adolescents will represent gender and minority distribution consistent with the Rochester metro/rural area demographic distribution. This study will be inclusive of all races, genders, and socioeconomic classes.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-10; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Cortical Excitability and Inhibition at Motor Cortex | Baseline
  Motor Threshold (MT) is a single-pulse TMS measure of cortical excitability. A higher MT indicates decreased cortical excitability. Intracortical Facilitation (ICF) is a paired-pulse TMS measure of cortical excitability. A higher ICF indicates increased cortical excitability. Cortical Silent Period (CSP) is a single-pulse TMS measure of cortical inhibition. Longer CSP durations indicate greater cortical inhibition. Intracortical Inhibition (ICI) is a paired pulse TMS measure of cortical inhibition. A lower ICI indicates increased cortical inhibition, and a higher ICI indicates decreased cortical inhibition.

SECONDARY OUTCOMES:
Glutamate Concentrations in the Motor Cortex and Anterior Cingulate Cortex | Baseline
  Glutamate concentrations will be measured with proton magnetic resonance imaging at 3T.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Croarkin, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Croarkin PE, Nakonezny PA, Husain MM, Port JD, Melton T, Kennard BD, Emslie GJ, Kozel FA, Daskalakis ZJ. Evidence for pretreatment LICI deficits among depressed children and adolescents with nonresponse to fluoxetine. Brain Stimul. 2014 Mar-Apr;7(2):243-51. doi: 10.1016/j.brs.2013.11.006. Epub 2013 Dec 3. PMID 24360599
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials